CLINICAL TRIAL: NCT03877510
Title: An Open-label Extension Study of the Safety and Clinical Utility of IPX203 in Parkinson's Disease Patients With Motor Fluctuations
Brief Title: Open Label Extension (OLE) Study of the Safety and Clinical Utility of IPX203 in Parkinson's Disease (PD) Participants With Motor Fluctuations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPX203-B16-03; 2018-002234-21 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: motor fluctuations; IPX203
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label IPX203 (Experimental): All participants received oral administration of extended-release capsules IPX203 dosing regimen that was determined at the end of the IPX203 dose conversion period of Study IPX203-B16-02 (NCT03670953) for nine months of open-label therapy. The dose and dosing frequency was determined by the investigator to achieve the optimal balance of efficacy and safety.
  Interventions: Drug: IPX203

INTERVENTIONS:
Drug: IPX203 — IPX203 extended release capsules

SUMMARY:
The purpose of this study is to evaluate the long-term safety and clinical utility of IPX203 in the treatment of participants with advanced Parkinson's disease (PD) who have motor fluctuations.

DETAILED DESCRIPTION:
This is a 9-month, multicenter open-label safety extension study. Participants who have successfully completed Study NCT03670953 [A Randomized Controlled Study to Compare the Safety and Efficacy of IPX203 with Immediate-Release (IR) Carbidopa-Levodopa (CD-LD) in Parkinson's Disease Patients with Motor Fluctuations] may have the opportunity to enroll in this open-label study.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed Study IPX203-B16-02
* Able to provide written informed consent prior to the conduct of any study-specific procedures.
* Female participants of childbearing potential must have a negative urine pregnancy test at the baseline visit (Visit 1).
* Agrees to use a medically acceptable method of contraception throughout the study and for 6 weeks after completing the study.

Exclusion Criteria:

* Intends to use any doses of Rytary® or Duopa™ during this study.
* Plans to use an investigational treatment other than IPX203 during the course of this study.
* Neurosurgical ablation treatment for PD is planned or anticipated during the study period. Implantation of a deep brain stimulator (DBS) for the treatment of PD is permitted during this study.
* Participants who, in the opinion of the clinical investigator, should not participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (98):
- United States (50):
  - Xenoscience, Inc (102), Phoenix, Arizona
  - St. Joseph's Hospital & Medical Center - Barrow Neurological Institute (156), Phoenix, Arizona
  - Clinical Trials, Inc (113), Little Rock, Arkansas
  - University of Arkansas for Medical Sciences (117), Little Rock, Arkansas
  - Keek School of Medicine of USC/ University of Southern California (106), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian (134), Newport Beach, California
  - SC3 Research-Pasadena (148), Pasadena, California
  - SC3 Research-Reseda (146), Reseda, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion (120), Aurora, Colorado
  - Rocky Mountain Movement Disorders (116), Englewood, Colorado
  - ChristianaCare Neurology Specialists (153), Newark, Delaware
  - JEM Research Institute (136), Atlantis, Florida
  - Visionary Investigators Network (168), Aventura, Florida
  - UHealth at Boca Raton (152), Boca Raton, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton (121), Boca Raton, Florida
  - Infinity Clinical Research LLC (104), Hollywood, Florida
  - University of Florida Health Science Center (129), Jacksonville, Florida
  - Neurology Associates, P.A. (125), Maitland, Florida
  - University of Miami (149), Miami, Florida
  - Medical Professional Clinical Research Center, Inc. (163), Miami, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida (131), Port Charlotte, Florida
  - Infinity Clinical Research, LLC (105), Sunrise, Florida
  - University of South Florida (114), Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology (174), West Palm Beach, Florida
  - Charter Research (166), Winter Park, Florida
  - Emory Brain Health Center (110), Atlanta, Georgia
  - NeuroStudies.net, LLC (155), Decatur, Georgia
  - Northwestern Medical Group Neurology Clinic (145), Chicago, Illinois
  - Central DuPage Hospital (151), Winfield, Illinois
  - Indiana University Health Neuroscience Center(164), Indianapolis, Indiana
  - University of Kansas Medical Center (118), Kansas City, Kansas
  - Quest Research Institute (103), Farmington Hills, Michigan
  - Henry Ford West Bloomfield Hospital(100), West Bloomfield, Michigan
  - Washington University (109), St Louis, Missouri
  - Roseman Medical Research Institute / Roseman Medical Group (154), Las Vegas, Nevada
  - Cleveland Clinic Lou Ruvo Center for Brain Health (142), Las Vegas, Nevada
  - Albany Medical College (139), Albany, New York
  - Ucgni (133), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center (123), Cleveland, Ohio
  - Cleveland Clinic(144), Cleveland, Ohio
  - University of Toledo, Gardner-McMaster Parkinson Center (122), Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma (115), Tulsa, Oklahoma
  - The Vanderbilt Clinic (158), Nashville, Tennessee
  - Neurology Consultants of Dallas, PA (108), Dallas, Texas
  - University of Texas Southwestern Medical Center (143), Dallas, Texas
  - Houston Methodist Neurological Institute/Movement Disorders Clinic (135), Houston, Texas
  - Inova Neurology- Fairfax (147), Fairfax, Virginia
  - VCU Health- Neuroscience Orthopaedic and Wellness Center(124), Henrico, Virginia
  - Booth Gardner Parkinson's Care Center (112), Kirkland, Washington
  - Inland Northwest Research (119), Spokane, Washington
- Czechia (6):
  - Fakultni nemocnice u sv. Anny v Brne, I. neurologicka klinika (704), Brno
  - NEUROHK. s.r.o. (701), Choceň
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Neurologicka klinika (702), Pardubice
  - CLINTRIAL s.r.o. (703), Prague
  - AXON Clinical. s.r.o. (700), Prague
  - Neurologicka ordinace FORBELI s.r.o. (706), Prague
- France (4):
  - CHU de Clermont-Ferrand-Hopital Gabriel Montpied (404), Clermont-Ferrand
  - CHU de Montpellier, Hopital Gui de Chauliac (405), Montpellier
  - Centre Hospitalier Universitaire de Nice (400), Nice
  - Centre d'lnvestigation Clinique 1436- CHU Purpan- Hopital Pierre Paul Riquet (403), Toulouse
- Germany (6):
  - Kliniken Beelitz GmbH, neurologisches Fachkrankenhaus fur Bewegungsstorungen/Parkinson (300), Beelitz-Heilstätten, Beelitz
  - St. Josef-Hospital, Universitatsklinik fur Neurologie Klinisches Forschungszentrum fur Neurodegeneration (301), Bochum, Gudrunstabe 56
  - Klinikum rechts der lsar der Technischen Universitat Munchen Klinik und Poliklinik fur Neurologie (303), München, Ismaningerstrabe
  - Dr. med. Reinhardt Ehret Neuroloqie Berlin Schlobstr. 29 (309), Berlin
  - Klinik Haag i. OB Geriatric Hospital Krankenhausstrabe 4 (305), Haag in Oberbayern
  - Gemeinschaftspraxis Dr. med. J. Springub/W. Schwarz, Studienzentrum Nordwest (306), Westerstede
- Italy (8):
  - Centro Ricerca Parkinson San Raffaele Cassino (601), Cassino, Frosinone
  - Università G. D'annunzio CeSi Met (604), Chieti, Italy/Chieti/Abbruzzo
  - Fondazione I st ituto Neurologico Nazionale "C. Mondino" (606), Pavia, Italy/Pavia/Lombardia
  - Azienda Ospedaliero-Universitaria Pisana (602), Pisa, Italy/Pisa/Toscana
  - IRCCS San Raffaele Pi sana (600), Roma, Italy/Roma/Lazio
  - Department of neuroscience, mental health and sensory system (NeSMOS), "Sapienza" University (603), Roma, Italy/Roma/Lazio
  - University of Rome Tor Vergata/Hospital Tor Vergata (605), Rome, Lazio
  - Department "G. F. Ingrassia" section of neuroscience - Policlinico "Vittorio Emanuele" (608), Catania, Sicily
- Poland (7):
  - Centrum Medyczne Neuromed (803), Bydgoszcz
  - Centrum Medyczne Linden (805), Krakow
  - Krakowska Akademia Neurologii Sp. Zo.o.(802), Krakow
  - NZOZ Neuromed M. i M. Nastaj Sp.p. (800), Lublin
  - NZOZ Neuro-Kard Ilkowski i Partnerzy Spolka Partnerska Lekarzy (801), Poznan
  - Neuro-Care Sp. z o.o. sp. k. (804), Siemianowice Śląskie
  - Centrum Medycme NeuroProtect (806), Warsaw
- Spain (14):
  - Hospital General Universitario de Elche (509), Elche, Alicante
  - Hospital Universitari General de Catalunya (504), Sant Cugat del Vallès, Barcelona
  - Hospital Universitari Mutua Terrassa (506), Terrassa, Barcelona
  - Policlinica Gipuzkoa, S.A (511), Donostia / San Sebastian, Gipuzkoa
  - Clinica Universidad de Navarra (512), Pamplona, Navarre
  - Hospital Universitario Quiron Dexeus (501), Barcelona
  - Germanes Hospitalaries Del Sagrat Cor De Jesus Hospital Sant Rafael (516), Barcelona
  - Hospital Universitario Vall d'Hebron (505), Barcelona
  - Hospital de Ia Santa Creu i Sant Pau (502), Barcelona
  - Hospital Universitario de Ia Princesa (508), Madrid
  - Hospital Universitario Ramon y Cajal (500), Madrid
  - Hospital Universitario Infanta Sofia(513), Madrid
  - Hospital Universitario Virgen del Rocio (503), Seville
  - Hospital Universitario y Politecnico La Fe Avenida Fernando Abril Martorell (515), Valencia
- United Kingdom (3):
  - Re:Cognition Health Ltd (205), Plymouth, Devon
  - Imperial College Healthcare NI-lS Trust (200), London
  - Re:Cognition Health Ltd (202), London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who successfully completed Study IPX203-B16-02 (NCT03670953) had the opportunity to enroll in the 9-month, open-label safety extension IPX203-B16-03 (NCT03877510) study. A total of 419 participants were enrolled.
Pre-assignment Details: Participants with Parkinson's Disease (PD) who were treated with stable regimens of carbidopa - levodopa (CD - LD) and had successfully completed previous IPX203-B16-02 study had the opportunity to enroll in this open-label study.
Period: Overall Study
Arm/Group | Open Label IPX203
Started | 419
Completed | 352
Not Completed | 67
Not completed — Death | 6
Not completed — Lost to Follow-up | 2
Not completed — Non-compliance with study drug | 2
Not completed — Lack of Efficacy | 14
Not completed — Adverse Event | 20
Not completed — Withdrawal by Subject | 22
Not completed — Miscellaneous | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were treated with the open-label study drug in the study.
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 419
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46
  Not Hispanic or Latino | 369
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 406
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical trial participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE was considered as treatment-emergent if the date of onset was on or after the date of the first open-label study drug administration in this Study IPX203-B16-03 and no later than 1 day after the last study drug dose in the study.
Time Frame: From first dose up to 1 day after last dose (Up to 9 months/Early Termination [ET])
Population: The Safety Analysis Set (SAS) included all participants who were treated with the open-label study drug in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 419
Participants | 221

2. Secondary Outcome: Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Total
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-260).
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: The Intent-to-Treat (ITT) Analysis Set included all participants who were treated with the open-label study drug in the study and had at least one post-baseline clinical utility assessment. "Overall Number of Participants Analyzed" included participants with available data at any timepoint. "Number Analyzed" included participants with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 409
  Baseline | 56.7 (28.64)
  Month 3: number analyzed (Participants) | 379
  Month 3 | 56.5 (30.14)
  Month 6: number analyzed (Participants) | 355
  Month 6 | 56.0 (28.92)
  Month 9/ET: number analyzed (Participants) | 393
  Month 9/ET | 59.0 (29.11)

3. Secondary Outcome: Change From Baseline in Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Total
Description: as for outcome 2
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 391
score on a scale | 2.7 (16.44)

4. Secondary Outcome: Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part I
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-260). Part I score ranges from 0 to 52. A higher score indicated more severe symptoms of PD.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with available data at any timepoint. "Number Analyzed" included participants with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 410
  Baseline | 9.9 (6.27)
  Month 3: number analyzed (Participants) | 390
  Month 3 | 10.6 (6.43)
  Month 6: number analyzed (Participants) | 362
  Month 6 | 10.7 (6.21)
  Month 9/ET: number analyzed (Participants) | 393
  Month 9/ET | 11.0 (6.72)

5. Secondary Outcome: Change From Baseline in Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part I
Description: as for outcome 4
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 392
score on a scale | 1.2 (4.56)

6. Secondary Outcome: Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part II
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-260). Part II score ranges from 0 to 52. A higher score indicated more severe symptoms of PD.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 409
  Baseline | 12.8 (7.83)
  Month 3: number analyzed (Participants) | 390
  Month 3 | 13.0 (7.96)
  Month 6: number analyzed (Participants) | 362
  Month 6 | 12.8 (7.69)
  Month 9/ET: number analyzed (Participants) | 393
  Month 9/ET | 13.6 (8.11)

7. Secondary Outcome: Change From Baseline in Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part II
Description: as for outcome 6
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 391
score on a scale | 0.9 (4.81)

8. Secondary Outcome: Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part III
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-260). Part III score ranges from 0 to 132. A higher score indicated more severe symptoms of PD.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 410
  Baseline | 27.5 (17.23)
  Month 3: number analyzed (Participants) | 379
  Month 3 | 26.8 (17.90)
  Month 6: number analyzed (Participants) | 357
  Month 6 | 26.6 (17.50)
  Month 9/ET: number analyzed (Participants) | 393
  Month 9/ET | 27.8 (16.79)

9. Secondary Outcome: Change From Baseline in Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part III
Description: as for outcome 8
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 392
score on a scale | 0.6 (11.29)

10. Secondary Outcome: Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part IV
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-260). Part IV score ranges from 0 to 24. A higher score indicated more severe symptoms of PD.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 410
  Baseline | 6.6 (2.96)
  Month 3: number analyzed (Participants) | 382
  Month 3 | 6.0 (3.15)
  Month 6: number analyzed (Participants) | 358
  Month 6 | 6.0 (3.08)
  Month 9/ET: number analyzed (Participants) | 393
  Month 9/ET | 6.6 (3.34)

11. Secondary Outcome: Change From Baseline in Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Part IV
Description: as for outcome 10
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 392
score on a scale | 0.0 (2.64)

12. Secondary Outcome: Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Sums of Part II and Part III
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 33 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-260). The scale range for Part II+III score is 0-184. A higher score indicated more severe symptoms of PD.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 409
  Baseline | 40.3 (23.09)
  Month 3: number analyzed (Participants) | 379
  Month 3 | 39.8 (24.15)
  Month 6: number analyzed (Participants) | 356
  Month 6 | 39.4 (23.24)
  Month 9/ET: number analyzed (Participants) | 393
  Month 9/ET | 41.5 (22.96)

13. Secondary Outcome: Change From Baseline in Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Sums of Part II and Part III
Description: as for outcome 12
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 391
score on a scale | 1.5 (13.66)

14. Secondary Outcome: Patient Global Impression of Severity (PGI-S)
Description: The PGI-S is a participant answered assessment rating Parkinson's disease severity on a scale of 1 to 7; 1-Normal, not at all ill, 2-Borderline ill, 3-Mildly ill, 4-Moderately ill, 5-Markedly ill, 6-Severely ill, 7-Extremely severely ill.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 409
  Baseline | 3.7 (1.02)
  Month 3: number analyzed (Participants) | 390
  Month 3 | 3.8 (1.00)
  Month 6: number analyzed (Participants) | 363
  Month 6 | 3.7 (0.99)
  Month 9/ET: number analyzed (Participants) | 393
  Month 9/ET | 3.8 (1.12)

15. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S)
Description: as for outcome 14
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 391
score on a scale | 0.0 (1.07)

16. Secondary Outcome: Percentage of Participants With a PGI-S ≥ 4 and PGI-S ≥ 5
Description: as for outcome 14
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: ITT population with available data was analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 409
Percentage of Participants
  Baseline PGI-S ≥ 4 | 64.5
  Baseline PGI-S ≥ 5 | 20.3
  Month 3 PGI-S ≥ 4: number analyzed (Participants) | 390
  Month 3 PGI-S ≥ 4 | 66.7
  Month 3 PGI-S ≥ 5: number analyzed (Participants) | 390
  Month 3 PGI-S ≥ 5 | 20.0
  Month 6 PGI-S ≥ 4: number analyzed (Participants) | 363
  Month 6 PGI-S ≥ 4 | 62.5
  Month 6 PGI-S ≥ 5: number analyzed (Participants) | 363
  Month 6 PGI-S ≥ 5 | 20.7
  Month 9/ET PGI-S ≥ 4: number analyzed (Participants) | 393
  Month 9/ET PGI-S ≥ 4 | 65.4
  Month 9/ET PGI-S ≥ 5: number analyzed (Participants) | 393
  Month 9/ET PGI-S ≥ 5 | 22.6

17. Secondary Outcome: Clinical Global Impression of Severity (CGI-S)
Description: The CGI-S is a clinician scale rating the severity of the participant's illness on a scale of 1 to 7; 1-Normal, not at all ill, 2-Borderline ill, 3-Mildly ill, 4-Moderately ill, 5-Markedly ill, 6-Severely ill, 7-Among the most extremely ill of participants.
Time Frame: Baseline, Month 3, Month 6, Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 409
  Baseline | 3.8 (0.87)
  Month 3: number analyzed (Participants) | 383
  Month 3 | 3.8 (0.92)
  Month 6: number analyzed (Participants) | 358
  Month 6 | 3.7 (0.87)
  Month 9/ET: number analyzed (Participants) | 392
  Month 9/ET | 3.8 (0.97)

18. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S)
Description: as for outcome 17
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 390
score on a scale | 0.0 (0.81)

19. Secondary Outcome: Percentage of Participants With a CGI-S ≥ 4 and CGI-S ≥ 5
Description: as for outcome 17
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: ITT population with available data was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 409
Percentage of participants
  Baseline CGI-S ≥ 4 | 66.7
  Baseline CGI-S ≥ 5 | 19.6
  Month 3 CGI-S ≥ 4: number analyzed (Participants) | 383
  Month 3 CGI-S ≥ 4 | 64.8
  Month 3 CGI-S ≥ 5: number analyzed (Participants) | 383
  Month 3 CGI-S ≥ 5 | 18.3
  Month 6 CGI-S ≥ 4: number analyzed (Participants) | 358
  Month 6 CGI-S ≥ 4 | 61.2
  Month 6 CGI-S ≥ 5: number analyzed (Participants) | 358
  Month 6 CGI-S ≥ 5 | 14.0
  Month 9/ET CGI-S ≥ 4: number analyzed (Participants) | 392
  Month 9/ET CGI-S ≥ 4 | 65.3
  Month 9/ET CGI-S ≥ 5: number analyzed (Participants) | 392
  Month 9/ET CGI-S ≥ 5 | 17.6

20. Secondary Outcome: 39-item Parkinson's Disease Questionnaire (PDQ-39): Total
Description: The PDQ-39 is a self-reported outcome of 39 questions relating to 8 domains: mobility (Questions 1-10), activities of daily living (ADL) (Questions 11-16), emotional well-being (Questions 17-22), stigma (Questions 23-26), social support (Questions 27-29), cognition (Questions 30-33), communication (Questions 34-36) and bodily discomfort (Questions 37-39). Each question is answered on a 5-point scale from 0 (Never) to 4 (Always / Cannot Do At All). Scores are calculated by summing the answers to the questions in the domain and converting to a scale from 0 to 100. Higher scores are associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 411
score on a scale
  Baseline: number analyzed (Participants) | 406
  Baseline | 41.7 (27.71)
  Month 3: number analyzed (Participants) | 392
  Month 3 | 42.7 (27.73)
  Month 6: number analyzed (Participants) | 364
  Month 6 | 42.8 (28.15)
  Month 9/ET: number analyzed (Participants) | 390
  Month 9/ET | 45.1 (29.45)

21. Secondary Outcome: Change From Baseline in PDQ-39: Total
Description: as for outcome 20
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 385
score on a scale | 4.4 (18.65)

22. Secondary Outcome: Parkinson Anxiety Scale (PAS): Total
Description: The PAS is a three part participant answered assessment. Part 1 has 5 questions measuring persistent anxiety. Each question ranges from 0 - not at all, or never to 4 severe, or nearly always. Best score is 0; worst score is 20. Part 2 has 4 questions measuring episodic anxiety. Each question ranges from 0 - never to 4 - nearly always. Best score is 0; worst score is 16. Part 3 has 3 questions measuring avoidance behavior. Each question ranges from 0, never to 4 nearly always. Best score is 0; worst score is 12. Totals for all three parts are summed and ranges from 0 to 48, higher scores are associated with the more severe symptoms.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 410
score on a scale
  Baseline: number analyzed (Participants) | 408
  Baseline | 10.4 (8.18)
  Month 3: number analyzed (Participants) | 390
  Month 3 | 10.3 (8.20)
  Month 6: number analyzed (Participants) | 365
  Month 6 | 10.3 (7.67)
  Month 9/ET: number analyzed (Participants) | 392
  Month 9/ET | 11.1 (8.57)

23. Secondary Outcome: Change From Baseline in Parkinson Anxiety Scale (PAS): Total
Description: as for outcome 22
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 389
score on a scale | 0.9 (6.41)

24. Secondary Outcome: Non-Motor Symptom Assessment Scale (NMSS) for Parkinson's Disease (PD): Total
Description: The NMSS assesses non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous. Severity symptoms are rated on a scale of 0-3 with 3 being most severe; and frequency on a scale of 1-4 with 4 being most frequent. Each question is answered with a severity and frequency rating which are then multiplied. The sum of the products gives the total score which ranges from 0 to 360 with a lower score more desirable than a higher score.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 407
  Baseline | 32.0 (28.95)
  Month 3: number analyzed (Participants) | 388
  Month 3 | 32.5 (28.49)
  Month 6: number analyzed (Participants) | 362
  Month 6 | 33.4 (29.19)
  Month 9/ET: number analyzed (Participants) | 392
  Month 9/ET | 35.3 (30.08)

25. Secondary Outcome: Change From Baseline in Non-Motor Symptom Assessment Scale (NMSS) for Parkinson's Disease (PD): Total
Description: as for outcome 24
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 389
score on a scale | 3.8 (22.33)

26. Secondary Outcome: Parkinson's Disease Sleep Scale-2 (PDSS-2) Total
Description: The PDSS-2 is a 15 question participant response scale measuring the severity of sleep disturbance. Three domains are defined: disturbed sleep (Questions 1-3, 8, 14), motor symptoms at night (Questions 4-6, 12, 13), PD symptoms at night (Questions 7, 9-11, 15). Each question is rated as very often to never on a scale of 0-4. The best overall score is 0; the worst overall score is 60.
Time Frame: Baseline, Month 3, Month 6, and Month 9/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 412
score on a scale
  Baseline: number analyzed (Participants) | 410
  Baseline | 16.6 (9.72)
  Month 3: number analyzed (Participants) | 389
  Month 3 | 15.8 (9.16)
  Month 6: number analyzed (Participants) | 363
  Month 6 | 16.1 (9.29)
  Month 9/ET: number analyzed (Participants) | 387
  Month 9/ET | 16.2 (9.28)

27. Secondary Outcome: Change From Baseline in Parkinson's Disease Sleep Scale-2 (PDSS-2):Total
Description: as for outcome 26
Time Frame: Baseline, Month 9/ET
Population: ITT population. "Overall Number of Participants Analyzed" included participants with Baseline and Month 9/ET data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 386
score on a scale | -0.1 (8.92)

28. Secondary Outcome: Treatment Satisfaction Assessment (TSA)
Description: The TSA is a participant answered assessment rating treatment satisfaction on a scale of 1 to 7; 1 = Very much dissatisfied being least satisfied and 7 = Very much satisfied.
Time Frame: Month 3, Month 6 and Month 9/ET
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 392
score on a scale
  Month 3 | 5.2 (1.25)
  Month 6: number analyzed (Participants) | 365
  Month 6 | 5.4 (1.19)
  Month 9/ET | 5.2 (1.39)

29. Secondary Outcome: Percentage of Participants With TSA Scores 5-7 (Satisfied) Versus Scores 1-4 (Dissatisfied or Neutral)
Description: as for outcome 28
Time Frame: Month 3, Month 6, and Month 9/ET
Population: ITT population with available data was analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Open Label IPX203
Number analyzed (Participants) | 392
Percentage of Participants
  Month 3: Percentage of TSA Scores 1-4 (Dissatisfied or Neutral) | 19.6
  Month 3: Percentage of TSA Scores 5-7 (Satisfied) | 80.4
  Month 6: Percentage of TSA Scores 1-4 (Dissatisfied or Neutral): number analyzed (Participants) | 365
  Month 6: Percentage of TSA Scores 1-4 (Dissatisfied or Neutral) | 15.6
  Month 6: Percentage of TSA Scores 5-7 (Satisfied): number analyzed (Participants) | 365
  Month 6: Percentage of TSA Scores 5-7 (Satisfied) | 84.4
  Month 9/ET: Percentage of TSA Scores 1-4 (Dissatisfied or Neutral) | 23.7
  Month 9/ET: Percentage of TSA Scores 5-7 (Satisfied) | 76.3

ADVERSE EVENTS:
Time Frame: From first dose up to 1 day after last dose (Up to 9 months/Early Termination [ET])
Arm/Group | Open Label IPX203
All-Cause Mortality (participants affected / at risk) | 6/419
Serious Adverse Events (participants affected / at risk) | 42/419
Other Adverse Events (participants affected / at risk) | 99/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label IPX203 (N=419)
Anemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Drowning (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 3
COVID-19 pneumonia (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Post procedural infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cauda equina syndrome (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Freezing phenomenon (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 3
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hypersexuality (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label IPX203 (N=419)
Constipation (Gastrointestinal disorders) | 11
COVID-19 (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 21
Fall (Injury, poisoning and procedural complications) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 15
Dyskinesia (Nervous system disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT03877510/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT03877510/SAP_001.pdf